CLINICAL TRIAL: NCT03150212
Title: Randomized Double Blind Placebo-controlled Clinical Study : Effect of IBSIUM on the Improvement of Gastro-intestinal Disorders Associated to the Irritable Bowel Syndrome (IBS) With C Phenotype (Predominant-constipation)
Brief Title: Effect of Saccharomyces Cerevisiae on the Improvement of Gastro-intestinal Disorders Associated to IBS With C Phenotype
Acronym: IBS-GO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-A01574-47
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saccharomyces cerevisiae CNCM I-3856 (Experimental)
  Interventions: Dietary Supplement: Saccharomyces cerevisiae CNCM I-3856
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces cerevisiae CNCM I-3856 — 2 capsules daily, just before the breakfast with a glass of water, during 8 weeks.
  Arms: Saccharomyces cerevisiae CNCM I-3856
Dietary Supplement: Placebo — 2 capsules daily, just before the breakfast with a glass of water, during 8 weeks.
  Arms: Placebo

SUMMARY:
The main objective is to assess the effect of an 8-week daily supplementation with IbSium® (probiotic yeast Saccharomyces cerevisiae CNCM I-3856) on the improvement gastro-intestinal disorders associated to the type C IBS (constipation predominant).

ELIGIBILITY:
Inclusion Criteria:

* Presenting IBS with predominant constipation according to the Rome IV criteria from at least 1 year and less than 10 years and without any possible doubt concerning confounding organic lesions (other organic pathologies having been excluded compliantly to the usual recommendations using differential diagnostic of chronic abdominal pain)

Rome IV:

A) Recurrent abdominal pain, with an average of at least 1 day a week within the last 3 months, and associated with 2 following criteria:

1. Related to defecation,
2. Associated with a change in stool frequency,
3. Associated with a change of the stools appearance.

B) Onset of the above symptoms at least 6 months before the diagnostic,

C) More than one-fourth (25%) of bowel movements with Bristol stool form types 1 or 2 and less than one-fourth (25%) of bowel movements with Bristol stool form types 6 or 7 (check during the last 14 days using the stools frequency questionnaire associated to the Bristol Stools Scale "BSS"),

* Score of abdominal pain/discomfort ≥ 2 and < 6 (using a 0 to 7 Likert point scale; daily average during the last 14 days verified at V1),
* For non-menopausal women: with the same efficient contraception method since at least 3 months before the start of the study, and accepting to maintain this program over the study (hormonal contraception, intrauterine device or surgical intervention). For menopausal women: with or without Hormone Replacement Therapy (HRT in place since less than 3 months before the start of the study are excluded) ,

Exclusion Criteria:

* Suffering from gastro-intestinal troubles other than IBS: lactose intolerance, Crohn disease, ulcerative colitis, celiac disease (gluten intolerance), symptomatic diverticulosis,
* Suffering from an immunodeficiency or affected by a severe or progressive disease (cardiac, pukmonary, hepatic, renal, hematologic, infectious or neoplastic),
* Suffering from a metabolic trouble affecting the intestinal transit function or the nutrients absorption like diabetes or unbalanced thyroid dysfunction,
* Currently under symptomatic drug treatment acting on the intestinal sensitivity or motility (laxatives, antispasmodics, anxiolytics, antidepressants, analgesics and NSAIDs are authorized if consumed for more than 3 months with a stable dosage and maintained during the study; opioïds and narcotic analgesics are forbidden), or dietary supplementation which according to the investigator should affect study results or stopped within a too short time window before the V1 randomization visit (less than 4 weeks for oral antibiotics, pre- or probiotics, less than 2 weeks for oral antifungal and anti-diarrheal if gastroenteritis),
* Refusing to stop the consumption of probiotics, prebiotics, or symbiotics under dietary supplement presentation or "health foods" (i.e. Lactibiane®, BION®, ultra yeast, kefir or food stuffs like ACTIMEL®, ACTIVIA® or other probiotics enriched dairy product etc.),
* Pregnant or lactating woman or intenting to become pregnant within 3 months ahead,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Abdominal pain/discomfort score rated with Likert scale (ranging from 0 to 7) | Week 5 to Week 8
  Total AUC W5-W8 (expressed in a.u./day.week) of abdominal pain/discomfort calculated using the mean daily score rated with Likert scale (ranging from 0 to 7) from week 5 to week 8 (included)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle METREAU, MD, Principal Investigator — Biofortis Mérieux NutriSciences; Arnaud BOURREILLE, Doctor, Principal Investigator — Service d'Hépatogastroentérologie - CHU Nantes; Pierre DESREUMAUX, Professor, Principal Investigator — Service de Gastroentérologie - Hôpital Huriez, CHU Lille
Locations (5):
- France (5):
  - General pratices, France
  - Eurofins Optimed, Gières
  - Créabio Rhône Alpes, Givors
  - Institut Pasteur de Lille, Lille
  - Biofortis Mérieux NutriSciences, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mourey F, Decherf A, Jeanne JF, Clement-Ziza M, Grisoni ML, Machuron F, Legrain-Raspaud S, Bourreille A, Desreumaux P. Saccharomyces cerevisiae I-3856 in irritable bowel syndrome with predominant constipation. World J Gastroenterol. 2022 Jun 14;28(22):2509-2522. doi: 10.3748/wjg.v28.i22.2509. PMID 35979259